CLINICAL TRIAL: NCT07273240
Title: The Effects of Physical Activity Program on Psychomotor and Psycho-Social Characteristics of Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Ayaz, Independent Researcher, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06.05.2022-376308; 06.05.2022-376308 (Other: Istanbul University-Cerrahpaşa)
Record Dates: First submitted 2025-11-16; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Children With Autism Spectrum Disorder
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Physical Activity Program
  Interventions: Other: Physical Activity
- control group (No Intervention): No intervention

INTERVENTIONS:
Other: Physical Activity — PAP was prepared for psychomotor (motor skills and physical fitness) and psychosocial (social skills and daily living skills) development areas based on the pre-test items of the data collection tools.
  Arms: experimental group

SUMMARY:
The aim of this study was to examine the effect of Physical Activity Program (PAP) on psychomotor and psychosocial characteristics of autistic children.

DETAILED DESCRIPTION:
The research group consisted of a total of 40 participants, 20 in the control group (CG) and 20 in the experimental group (EG), aged between 8-12 years. EG participated in the PAP for 60 minutes a day, 3 days a week for 10 weeks. Gilliam Autistic Disorder Rating Scale-2, Bruininks-Oseretsky motor competence test-2 short form (BOT-2 SF), Eurofit Test Battery, Pediatric Quality of Life Form and Social Skills Rating System Parent Form were used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Recognized ASD
* Between 8 and 12 years of age
* Attending a special education school
* No impairment of vision, hearing, or acceleration
* No health problems that would prevent economic activity
* Not participating in any sports
* Updated procedures by the parent.

Exclusion Criteria:

* Family withdrawal from the study
* Failure to participate in pre-tests or post-tests
* Absence from the program for more than two weeks

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
The effect of physical activity on psychomotor characteristics | 10-week physical activity program
  Outcome Name: Change in gross motor skills Description: Measured using the Bruininks-Oseretsky Test of Motor Proficiency (BOT-2), total and subscale scores.

SECONDARY OUTCOMES:
The effect of physical activity on psychomotor characteristics | 10-week physical activity program
  Outcome Name: Change in gross motor skills Description: Measured using total and subscale scores using the Eurofit Test Battery.

OTHER OUTCOMES:
The effect of physical activity on psychososyal characteristics | 10-week physical activity program
  Outcome Name: Change in psychosocial skills Description: Psychosocial characteristics were measured using the Gilliam Autism Disorder Rating Scale-2.
The effect of physical activity on psychosocial characteristics | 10-week physical activity program
  Outcome Name: Change in gross psychosocial skills Description: Psychosocial characteristics were measured using the Pediatric Quality of Life Form.
The effect of physical activity on psychosocial characteristics | 10-week physical activity program
  Outcome Name: Change in gross psychosocial skills Description: Psychosocial characteristics were measured using the Social Skills Rating System Parent Form

CONTACTS AND LOCATIONS:
Overall Officials: Dilara F Özer, Prof. Dr., Study Director — İstanbul Bilgi University; Gülsüm H Özcan, Dr., Study Chair — İstanbul University Cerrahpaşa
Locations (1):
- Izmit Special Education Practice School, Derince Special Education Practice School, Golcuk Ozdebir Special Education Practice Center, Kartepe Special Education Practice School, Izmit, Kocaeli 41500, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPDs that form the basis of a publication's results
Supporting Information: Study Protocol
Time Frame: Individual participant data and supporting documentation will be made available 6 months after the main results are published and will remain available for 5 years.
Access Criteria: Individual participant data and supporting documentation will be made available to qualified researchers upon reasonable request. Access will be granted for scientific research proposals that have received ethics committee approval, and researchers will be required to sign an access agreement outlining data use and confidentiality terms.

REFERENCES:
- See also: Related Info — https://www.iuc.edu.tr/

DOCUMENTS (3):
  • Study Protocol (2022-04-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT07273240/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT07273240/SAP_001.pdf
  • Informed Consent Form (2022-04-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT07273240/ICF_002.pdf